CLINICAL TRIAL: NCT00789399
Title: A Study of the Efficacy of Preventive Dosing of Fondaparinux Sodium Versus Placebo for the Prevention of Venous Thromboembolism (VTE) in Patients Undergoing Coronary Bypass Surgery Receiving Routine Mechanical Prophylaxis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator moved to another region of the country
Sponsor: Prairie Education and Research Cooperative (Industry)
Collaborators: American College of Phlebology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00508826
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Deep Vein Thrombosis; Coronary Artery Bypass Surgery; Venous Thromboembolism
Keywords: deep vein thrombosis; coronary artery bypass surgery; Venous thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism | interventions — Fondaparinux

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fondaparinux (Active Comparator): Patients will receive a 2.5 mg dose of Fondaparinux subcutaneously for a total of 7 days post CABG
  Interventions: Drug: Fondaparinux
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fondaparinux — Patients will receive a 2.5 mg dose of Fondaparinux subcutaneously for a total of 7 days post CABG
  Other Names: DVT; CABG
  Arms: Fondaparinux
Other: Placebo — subcutaneous equivolume isotonic saline
  Other Names: DVT; CABG
  Arms: Placebo

SUMMARY:
This trial is a prospective, single-center Phase II randomized study to demonstrate the superior efficacy of Fondaparinux Sodium subcutaneous injections in patients undergoing CABG surgery (isolated and redo isolated) versus treatment with placebo. All consecutive patients scheduled for CABG surgery that meet the general inclusion and none of the exclusion criteria will be considered for enrollment in the study.

Consecutive patients will be randomized on the day of admission prior to their CABG surgery into one of two groups. One group will be randomized to the placebo while the second group will receive 2.5 mg Fondaparinux Sodium injections. Both groups will receive routine mechanical prophylaxis as determined by the treating physicians. Group randomized to receive Fondaparinux Sodium will receive a 2.5 mg SQ daily drug dose starting 12 +/- 2 hours post-wound closure or the following day in the morning (at the discretion of the cardiothoracic surgeon). The second dose would be administered 24 hours later and the dosing will then be once a day. The group randomized to placebo will receive subcutaneous equivolume isotonic saline at the same time points described above.

Patients randomized will receive a 2.5 mg dose of Fondaparinux Sodium or placebo subcutaneously for a total of 3-9 days post CABG with day 1 being the day of surgery. The drug will be discontinued if the patient is discharged before day 9. If the patient stays for more than 9 days inside hospital, a duplex would be obtained per protocol and further DVT prevention measures would be instituted per the discretion of treating physician.

Patients will be assessed daily while hospitalized for any symptoms and adverse reactions and will undergo laboratory testing (CBC, PT/INR, PTT and UA) as specified in the protocol. Post-op day 3-9(no later than 2 days after the last preventive drug dose) patients will undergo the protocol specific lower limb venous duplex scan and earlier if symptomatic. Patients will also be contacted (phone/office visit) for follow-up 25-35 days post CABG to assess for signs or symptoms of deep venous thrombosis or thromboembolism and for any potential complications.

DETAILED DESCRIPTION:
Background Information

Venous thromboembolism (VTE) following coronary artery bypass graft (CABG) surgery is a formidable risk in view of various predisposing factors including restriction of activity, history of myocardial infarctions in such patients, presence of multiple predisposing baseline demographic characteristics and risk factors including advanced age and smoking. The reported incidence of asymptomatic deep vein thrombosis (DVT) using duplex ultrasound (DUS) is significant and varies from 16 to 48%, most of the thrombi being calf vein. (1,2,3) The incidence of symptomatic VTE based chiefly on retrospective data ranges from 0.5 to 3.9% for VTE, 0.3 to 0.5% for DVT, 0.2 to 3.9% for PE, and 0.06 to 0.7% for fatal PE. (2-10)The absolute number of affected patients may be significant since the number of such procedures performed every year in the US alone is huge. According to the American Heart Association's Heart Disease and Stroke Statistics - 2008 Update, 469,000 surgical revascularizations were done in the US in 2005.

The benefits of thromboprophylaxis in medically ill patients including those with congestive heart failure have been well demonstrated with up to 60% reduction in VTE risk. (11) The patients who undergo CABG have similar risk profiles and hence should be evaluated with pharmacokinetic thromboprophylacic strategy.

In CABG patients, the American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition), 2008, (12) does recommend routine prophylaxis with low molecular weight heparin (LMWH), low dose unfractionated heparin (LDUH), or optimally used bilateral graduated compression stockings (GCS) or intermittent pneumatic compression (IPC). The guidelines are based on moderate to low quality evidence and the strength of these recommendations is weak as there have been no randomized controlled trials.

Rationale In CABG patients, the American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition), 2008,(12) recommend routine prophylaxis with LMWH, LDUH, or optimally used bilateral GCS or IPC. The guidelines are based on moderate to low quality evidence and the strength of the recommendation is weak as there have been no randomized controlled trials. Optimally used stockings may not be applicable to many CABG patients because of saphenous vein harvesting and hence pharmacologic means are preferable.

Fondaparinux is a pentasaccharide with an efficacy and safeties shown to be equal to or better than LMWH and thus may be a preferred agent for VTE prophylaxis. (13-18)

OBJECTIVES The primary goal of this study is to demonstrate the superiority of Fondaparinux Sodium over placebo for the prevention of VTE in Patients undergoing Coronary Bypass Graft Surgery (CABG).

Primary Efficacy Endpoint:

• Cumulative incidence of all VTE (defined as symptomatic and asymptomatic deep-vein thrombosis, fatal and non-fatal pulmonary embolism, or both) up to day 11

Secondary Efficacy Endpoints:

• Primary efficacy end-point and VTE up to day 35

Primary Safety Endpoints:

• Major bleeding event up to day 11

Secondary Safety Endpoints:

* Cumulative major and minor bleeding event up to day 11
* Deaths, requirement of transfusions and other adverse events up to day 35

STUDY DESIGN This trial is a phase II, prospective, single-center, assessor and patient-blinded, placebo controlled, randomized study to demonstrate the superior thromboprophylactic efficacy of Fondaparinux Sodium subcutaneous injections in patients undergoing CABG surgery versus placebo.

OBJECTIVES The primary efficacy objectives include an assessment of the cumulative rate of all VTE (defined as DVT or fatal or non-fatal pulmonary embolism or both) up to 11 days post CABG. The primary safety objectives include the assessment of the frequency and occurrence of all major bleeding events post-operatively up to day 3-11. Finally, the secondary efficacy objective will include cumulative VTE events and assessment of the components of VTE while the secondary safety objective will include an assessment of the frequency of non-major bleeding events up to day 3-11 as well as all cause deaths, need for transfusion and other monitored adverse events till day 35. The inclusion of safety is mainly for descriptive purposes because the study is not be powered for safety end points.

The safety and efficacy endpoints will determine Fondaparinux Sodium's ability over placebo to prevent VTE while assessing the bleeding risk in this study population. A randomized control is needed because a head to head comparison of Fondaparinux Sodium and placebo is being planned.

Approximate time to complete study enrollment is 2 years. This estimation is based on the number of subjects needed for the study and the rate of CABG surgery performed at the institution.

ELIGIBILITY:
Subject Inclusion Criteria In order to be enrolled in the study, subjects must meet all of the inclusion criteria as listed below.

1. Consecutive patients undergoing isolated or redo isolated CABG
2. Patients must provide written informed consent
3. Patients must agree to comply with study procedures for the entire length of the study.
4. Must be 18 years old or greater.

Subject Exclusion Criteria Any subject that meets any of the exclusion criteria listed below at baseline will be excluded from study participation.

1. Patients with medical history that requires chronic anticoagulation with unfractionated heparin or coumadin or LMWH or heparinoids (i.e. previous DVT, pulmonary embolism, atrial fibrillation, heart valve replacement)
2. Patients with contraindications to anticoagulation (coagulopathy e.g, INR>/=1.5, generalized bleeding disorders, peptic ulcer disease, hemorrhagic or ischemic stroke, etc within last 3 months)
3. Patients who are unable to undergo a doppler ultrasound of the lower extremities
4. Renal insufficiency (creatinine clearance < 30 mL/min)
5. Patients who have a body weight < 50 kg
6. Patients receiving continuous (indwelling) epidural
7. Physician diagnosed acute or chronic hepatic failure
8. Pregnancy
9. Patients with life expectancy < 6 months
10. Platelet count below 100,000/ mm-3
11. History of documented VTE within last 3 months.
12. Acute bacterial endocarditis
13. Cerebral metastasis or abscess
14. Inability to consent
15. Refusal by treating physician

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-11-19 (Actual); Primary Completion 2013-09-21 (Actual); Study Completion 2013-09-21 (Actual)

REFERENCES:
- [Derived] Kolluri R, Plessa AL, Sanders MC, Singh NK, Lucore C. A randomized study of the safety and efficacy of fondaparinux versus placebo in the prevention of venous thromboembolism after coronary artery bypass graft surgery. Am Heart J. 2016 Jan;171(1):1-6. doi: 10.1016/j.ahj.2015.10.013. Epub 2015 Oct 21. PMID 26699594

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fondaparinux | Placebo
Started | 41 | 37
Completed | 39 | 37
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fondaparinux | Placebo | Total
Number analyzed (Participants) | 41 | 37 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (8.9) | 62 (8.9) | 63.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 30 | 27 | 57
Region of Enrollment [Number; unit: participants]
  United States | 41 | 37 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolisms and/or Major Hemorrhages to Day 11
Description: there were 2 events; one in placebo group and one in fondaparinux group
Time Frame: 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fondaparinux | Placebo
Number analyzed (Participants) | 41 | 37
Participants | 1 | 1

2. Secondary Outcome: Number of Participants With a Venous Thromboembolisms to 35 Days
Time Frame: 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fondaparinux | Placebo
Number analyzed (Participants) | 41 | 37
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 year follow up
Groups:
- Fondaparinux Subjects: pts received fondaparinux
- Placebo Subjects: patients received placebo
Arm/Group | Fondaparinux Subjects | Placebo Subjects
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/37
Serious Adverse Events (participants affected / at risk) | 34/41 | 18/37
Other Adverse Events (participants affected / at risk) | 19/41 | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fondaparinux Subjects (N=41) | Placebo Subjects (N=37)
DVT (Vascular disorders) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
CHF (Cardiac disorders) | 10 (10) | 4 (4)
cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
cardiac arrhythmia (Cardiac disorders) | 7 (7) | 2 (2)
Afib/Aflutter (Cardiac disorders) | 11 (11) | 4 (4)
Other Cardiac (Cardiac disorders) | 7 (8) | 3 (3)
Resp Arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Other Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Surgical Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Other Infections (Infections and infestations) | 4 (4) | 1 (1)
Other Neurological (Nervous system disorders) | 1 (1) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 2 (2) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Other GI (Gastrointestinal disorders) | 5 (5) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
other (General disorders) | 13 (16) | 8 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fondaparinux Subjects (N=41) | Placebo Subjects (N=37)
Other, Pulmonary (Respiratory, thoracic and mediastinal disorders) | 14 (25) | 14 (26)
Other, Cardiac (Cardiac disorders) | 1 (1) | 4 (4)
Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
surgical site infection (Infections and infestations) | 1 (1) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
other (General disorders) | 5 (7) | 7 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No